CLINICAL TRIAL: NCT02322164
Title: Psychophysical Correlates of Pain Reduction by Topical Analgesic Compounds
Status: Completed | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150048; 15-AT-0048
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2018-07-02

CONDITIONS: Healthy Volunteers
Keywords: Skin; TEMPERATURE; Placebo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Researchers are studying a topical (skin) cream that reduces pain. This is called an analgesic cream. They want to try a new test to better measure how well it works. Heat will be applied to the participants arms and they will judge the intensity of the temperatures. Researchers will compare the pain reduction from this cream to other pain relief treatments.

Objective:

- To better measure the effects of a pain-relieving (analgesic) cream.

Eligibility:

- Healthy volunteers ages 18 50.

Design:

* There will be 2 study sessions.
* Session 1 will be about 1.5 hours.

  * Participants will be screened with physical exam and urine drug test. They will answer medical and psychological questions.
  * Participants will have sensory testing.
* A moisturizer will be put on their arms. A heating device will be placed on their arms. It gives heat pulses of about 2 seconds each. Some are warm and some are very hot. Participants will say how strong each pulse is. They can move away if it gets painful.
* Then the pain-relieving cream will be put on one arm. The moisturizer will be put on the other. Participants will get more pulses and rate them. They will also get pairs of pulses and compare them.
* Some participants will return for session 2 for 1 hour. They will receive similar sensory testing as in session 1.

DETAILED DESCRIPTION:
This study uses a new testing design to evaluate pain reduction from a pain-relieving cream. Sequences of heat stimuli will be applied to the participants arms and participants will be asked to judge the intensity of the temperatures they perceive. There are two study sessions. Session 1 involves eligibility screening and baseline sensory testing with and without the analgesic (pain-relieving) cream. Session 2 involves more sensory testing with the analgesic cream. The study population is 40 healthy volunteers aged 18 to 50.

ELIGIBILITY:
* INCLUSION CRITERIA:

You may be eligible to participate in this research study if you are:

1. Between 18 and 50 years old.
2. Fluent in English.
3. Able to understand the procedures described in this document and give your written consent.

EXCLUSION CRITERIA:

You may not be eligible to participate in this research study if you:

1. Cannot complete the required procedures and tests in the study
2. Used recreational drugs within the past six months
3. Are in the third trimester of pregnancy
4. Have a major medical condition or major medical history event that could affect touch and pain
5. Have a medical condition that might affect touch and pain (e.g. Raynaud s Disease, peripheral neuropathy, or circulatory disorder)
6. Have chronic pain or a history or chronic pain
7. Have allergies to topical treatments
8. Have a dermatological condition such as scars or burns, or have had a tattoo on your forearms within the previous four weeks that might influence touch or pain
9. Had a recent or permanent injury of upper limbs or amputation or use a prosthetic limb
10. Have participated in related NIH protocols (we will determine this)
11. Used non-steroidal anti-inflammatory drugs (NSAIDS, e.g. aspirin, ibuprofen), acetaminophen, or sumatriptan within 3 days of testing (brand names include Advil, Tylenol, and Imitrex)
12. Used narcotics (e.g. opioids, oxycodone) or pseudo narcotics (e.g. tramadol, tapentadol) within one week of testing (brand names include Percocet and Ultram)
13. Use centrally acting medications like anticonvulsants (e.g. gabapentin, pregabalin), antidepressants (e.g. fluoxetine, duloxetine), antipsychotics (e.g. chlorpromazine, prochlorperazine), or anxiolytics (e.g. clonazepam, alprazolam) (Brand names include Neurontin, Lyrica, Prozac, Cymbalta, and Xanax)
14. Use tobacco daily or used tobacco within 24 hours of testing
15. Used topical pain-relieving creams in the testing area (e.g. methylsalicylate, capsaicin) within 24 hours of testing (Brand names include IcyHot and BenGay)
16. Cannot schedule two sessions within two weeks
17. Have consumed caffeine before 2 hours of testing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-12-19; Primary Completion 2017-09-21 (Actual); Study Completion 2018-07-02 (Actual)

PRIMARY OUTCOMES:
Thermal sensory discrimination | One time point

CONTACTS AND LOCATIONS:
Overall Officials: Mary C Bushnell, Ph.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States